CLINICAL TRIAL: NCT00161889
Title: Follow-up Study to Investigate the Safety and Immunogenicity of a Third Vaccination With Three Different Antigen Concentrations of FSME IMMUN NEW in Children Aged 6 to 16 Years
Brief Title: FSME IMMUN NEW Follow-up to Study 205 in Children Aged 6 to 16 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 207
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-borne
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated)

SUMMARY:
The purpose of this study is to investigate the safety and immunogenicity of the third vaccination with one of three different concentrations of a TBE vaccine in all volunteers who completed two vaccinations in one of the three treatment groups of Baxter study 205 (safety and immunogenicity of two vaccinations with FSME IMMUN NEW in healthy volunteers aged 6 to 16 years).

ELIGIBILITY:
Inclusion criteria:

All volunteers who participated in Baxter study 205 and received two vaccinations will be invited to participate. Male and female children will be eligible for participation in this study if:

* They received two vaccinations with one of the three different dosages of FSME IMMUN NEW during the course of Baxter study 205
* They and/or their legal guardian understand the nature of the study, agree to its provisions and give written informed consent

Exclusion Criteria:

There are no specific exclusion criteria for this study entry. However volunteers will be assessed for eligibility to receive a third vaccination.

Volunteers will be excluded from vaccination and consecutive visits in this study if they:

* Are not clinically healthy, (i. e. the physician would have reservations vaccinating with FSME IMMUN NEW outside the scope of a clinical trial)
* Have already been administered a third TBE vaccination elsewhere after the two vaccinations in Baxter study 205
* Have had an allergic reaction to one of the components of the vaccine since the last vaccination in Baxter study 205
* Suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids, chemotherapeutics) that can be expected to influence immunological functions
* Have received banked human blood or immunoglobulins within one month of study entry
* Are known to be HIV positive (a special HIV test is not required for the purpose of the study) since the last visit of Baxter study 205
* Have had a vaccination against yellow fever and / or Japanese B-encephalitis since the last visit in Baxter study 205
* Had received an investigational new drug within 6 weeks prior to study start
* If female and capable of bearing children - have a positive pregnancy test at the first medical examination

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 615
Dates: Start 2002-02; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (19):
- Germany (19):
  - Neuschwanstein Strasse 5, Augsburg
  - Marktplatz 33, Bad Saulgau
  - Hauptstrasse 9, Bietigheim-Bissingen
  - Salzgasse 11, Calw
  - Mohrenstrasse 8, Coburg
  - Bahnhofstrasse 1, Elzach
  - Rheinstrasse 1a, Ettenheim
  - Peter-Seifert Strasse 5, Gersfeld
  - Solothumer Strasse 2, Heilbronn
  - Hauptstrasse 240, Kehl
  - Schwarzwald Strasse 20, Kirchzarten
  - Altoettinger Strasse 3, Landsberg
  - Rastatter Strasse 7, Mannheim-Secken
  - Wilhelmstrasse 25, Metzingen
  - Dohmbuehler Strasse 8, Nuremberg
  - Wilhelmstrasse 7, Offenburg
  - Berneckstrasse 19, Schramberg
  - Hauptstrasse 11, Tegernsee
  - Broner Platz 6, Weingarten